CLINICAL TRIAL: NCT03867864
Title: Hao-Yuan Chang, Assistant Professor, School of Nursing, National Taiwan University
Brief Title: Effects of Aromatherapy on the Headache and Service Quality Among Nurses Working in Critical Care Nurses Units.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 201710020RINA
Record Dates: First submitted 2019-03-06; First posted 2019-03-08 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-02

CONDITIONS: Headache, Migraine; Quality of Life
Keywords: Headache; Migraine; Disability; Quality of life; Nurse; Aromatherapy; Essential oils; Missed care
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — WASH protein, Drosophila

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A participants will wear the necklace with essential oil for the first 4 weeks except take a shower or get to sleep. The participants will stop wearing the necklace for one week (the fifth week) for washout period, and then wear the necklace without essential oil for last 4 weeks (the sixth to ninth weeks).
  Interventions: Device: Necklace with essential oil for the first 4 weeks; Other: Washout; Device: Necklace without essential oil for last 4 weeks
- Group B (Other): The group B will wear the necklace without essential oil for the first 4 weeks except take a shower or get to sleep. The participants will stop wearing the necklace for one week (the fifth week) for washout period, and then wear the necklace with essential oil for last 4 weeks (the sixth to ninth weeks).
  Interventions: Device: Necklace without essential oil for the first 4 weeks; Other: Washout; Device: Necklace with essential oil for last 4 weeks

INTERVENTIONS:
Device: Necklace with essential oil for the first 4 weeks — The necklaces contain essential oil.
  Arms: Group A
Device: Necklace without essential oil for the first 4 weeks — The necklaces do not contain essential oil.
  Arms: Group B
Other: Washout — Washout (do not wear the necklace) for one week for two groups, then two groups cross-over.
Device: Necklace with essential oil for last 4 weeks — The necklaces contain essential oil.
  Arms: Group B
Device: Necklace without essential oil for last 4 weeks — The necklaces do not contain essential oil.
  Arms: Group A

SUMMARY:
Background: Our pilot study showed that the prevalence of headaches is 43.5% among nurses working in critical care units in a medical center in Taiwan. In the pilot study, 70% nurses with headache are willing to participate in this intervention study with essential oil. The effect of aromatherapy (essential oils through smelling) is convenient for nurses but still lacks strong evidences regarding relieving headaches.

Purpose: Thus, in this intervention study, we will examine whether the necklace with essential oil can (1) improve the pain intensity and frequency of headache; (2) reduce the score of headache disability inventory (HDI) and (3) improve the nurses' quality of life and care quality.

Method: Cluster randomized control trial from 16 critical care units at a medical center in Taiwan. The International Classification of Headache Disorders (ICHD, 3rd edition) was used to identify the headache type as "migraine" or "tension-type headache." We will recruit the nurses from 16 critical care units who has migraine or tension-type headache and cluster random assign (according to the ward unit) to group A and B. The intervention of necklace with essential oil will use to compare with the other group. According to power analysis and possible attrition rate, 103 nurses will be recruited. All participants will be asked to complete self-administrated questionnaires, including headache information questions, headache disability inventory (HDI), Migraine Specific Quality of Life Questionnaire version 2.1 (MSQv2.1), Copenhagen burnout inventory (CBI), Service Quality Scale (SERVQUAL), Intention to leave inventory (ITL), Depression, Anxiety and Stress Scale (DASS-21), Tasks Undone-13 (TU-13). The quantitative data will analyze by percentage, mean, standard deviation, chi-square test, and generalized estimating equation (GEE).

Expected outcomes and future implications: The aromatherapy (necklace with essential oil) can reduce the pain intensity, frequency, disability of headaches, as well as enhance nurses' quality of life and care quality.

DETAILED DESCRIPTION:
This study adopts an experimental design with cluster randomization based on the ward unit. Eligible subjects are diagnosed migraine or tension-type headache nurses who are working in the critical care units and also have nurse license. Before conducting this study, the study has been approved by the institutional review board (IRB). The researcher (co-PI) and research assistances will approach potential participants during the ward meeting and invite them to participate in the study. Potential participants would be informed of the study purposes and interventions process, and be assessed and confirmed their type of headache. After completing the written-informed consent, the interventions will be arranged. In order to control the quality of data collection, PI and co-PI have trained the research assistants. Research training included standardized research process and ethical concerns about collection of research data, methods of approaching eligible subjects, interviewing techniques of data collection.

ELIGIBILITY:
Inclusion Criteria:

* Registered nurses, working in intensive care units (ICU) or department of emergency (ED).
* The frequency of headaches more than three times per month.
* The type of headache is migraine or frequent episodic tension-type headache, which is defined by the Headache Classification Committee of the International Headache Society. If the symptoms of a headache cannot be defined, the investigator will refer the potential participant to a neurologist for further diagnosis.

Exclusion Criteria:

* Current user of other kinds of essential oils (e.g., the external application on skin, sniffing), and do not willing to temporarily suspend for nine weeks.
* Having sensitive responses to the essential oil.
* Pregnancy or preparing for pregnancy.
* Breastfeeding.
* The type of headache was neither migraine nor frequent episodic tension-type headache after diagnosed by the neurologist.
* With hepatic or renal diseases.
* taking medicine for long-term (such as Aspirin, anti-coagulant, medication for mental disorders, contraceptives, etc.).

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Estimated)
Dates: Start 2019-03-15 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of Headache Diary | The participants will be assessed among pre-test week 1 (T1) and persistent to fill out the headache diary every day for 9 weeks (totally 63 days)
  The Headache Diary measured the participants to record the condition of headache with 12 items. The investigators will analyzed the intensity, frequency, duration, location, quality, symptoms, time and medicine use, and the duration (hours) of wearing the necklace with essential oil. At the meanwhile, we also collect the perceived busy level of the work day to control the association between the workload and headache. Thus, the participants have to write the diary everyday for 9 weeks and we will remind them by the text. The diary also mixes in the short-form McGill pain questionnaire (SF-MPQ) that was developed by Melzack in 1975 and revised in 1987 and it developed from the different type of headache depending on the pain intensity and quality (Melzack, 1975). The investigators simplified the contents and transfer to code so that the participants can easily fill out the diary every day.
Changes of Headache Disability Inventory (HDI) | The participants will be assessed among pre-test week 1 (T1), week 5 (T2) and week 10 (T3)
  The Headache Disability Inventory (HDI) measured the burden caused by chronic headaches with 27 items (French et al., 2000). Each item scored from 1 to 3 (1= always happened; 3 = never happened). The higher score indicated the higher impacts of headache on emotional function and daily life.
Changes of Migraine Specific Quality of Life Questionnaire version 2.1 (MSQv2.1) | The participants will be assessed among pre-test week 1 (T1), week 5 (T2) and week 10 (T3)
  The Migraine Specific Quality of Life Questionnaire version 2.1 (MSQv2.1) measured the quality of life of migraine and headache patients, including the function, limitation, burden and impacts of the migraine with 14 items (Bagley et al., 2011). Each item was scored from 1 to 6 (1= always happened; 6 = never happened). The higher score indicated the higher impact of headache on quality of life. Cronbach's alphas are 0.79-0.85 (Bagley et al., 2011).
Changes of Copenhagen Burnout Inventory (CBI) | The participants will be assessed among pre-test week 1 (T1), week 5 (T2) and week 10 (T3)
  The Copenhagen Burnout Inventory (CBI) measured occupational burnout with 21 items (Yah et al, 2008). The questionnaire is including subscales-personal burnout, work-related burnout, client-related burnout, and over-commitment to work. Each item scored from 1 to 5 (1= never happened, 5 = always happened). The higher scores indicated the stronger work burnout. Cronbach's alphas are 0.89-0.95 (Yang et al, 2014).
Changes of Service Quality Scale (SERVQUAL) | The participants will be assessed among pre-test week 1 (T1), week 5 (T2) and week 10 (T3)
  The Service Quality Scale (SERVQUAL) measured the care quality of nurses in the hospital, including the four domains: trustworthiness, responsiveness, promise and empathy with 28 Likert's scale items (Teng et al., 2007). Each item scored from 1 to 5 (1= strongly disagree; 5 = strongly agree). The higher score indicated the higher confidence on their care quality.
Changes of Intention to Leave Inventory (ITL) | The participants will be assessed among pre-test week 1 (T1), week 5 (T2) and week 10 (T3)
  The Intention to Leave Inventory (ITL) measured the intention to leave the organization and their future career plan with 7 Likert's scale items (Teng, Shyu, & Chang, 2007). Each item scored from 1 to 7 (1= strongly disagree; 7 = strongly agree). The higher score indicated the higher strongly intention to leave the organization.
Changes of Depression, Anxiety and Stress Scale (DASS-21) | The participants will be assessed among pre-test week 1 (T1), week 5 (T2) and week 10 (T3)
  The Depression, Anxiety and Stress Scale (DASS-21) measured the level of depression, anxiety and stress during the past week recently by 21 items (Moussa, 2001). Each item scored from 1 to 4 (1= strongly disagree; 4 = strongly agree). The higher score indicated more frequency of feeling depression, anxiety and stress (Lovibond & Lovibond, 2004). Cronbach's alphas were 0.87-0.94 (Black et al., 2015).
Demographic and Headache Information Questionnaire | The participants will be assessed at pre-test week 1 (T1)
  The Demographic Questionnaire included the birth date, sex, marital status, amenorrhea, education, unit, working years and rank. Although the necklace's colors are distributed randomly, considering the color may also affect the participants 'mood or the condition of headache, therefore, The investigators also survey the subject's preference of color to control the potential effect. The Headache Information Questionnaire was modified from the International Classification of Headache Disorders (ICHD, 3rd edition) to identify the headache type as "migraine" or "tension-type headache. Items included pain intensity, frequency, onset of the times, symptoms, locations, etc.
Tasks Undone-13 | The participants will be assessed among pre-test week 1 (T1), week 5 (T2) and week 10 (T3)
  The tasks undone-13 measured the missed care with 13 items (Aiken et al; Ball et al., 2013; Schubert, 2007). Each item scored from 0 to 1 (0 = left done, 1 = done and NA= not applicable) The higher score indicated the volume of care left done. Cronbach's alpha = 0.73 (Lucero et al., 2009) and content validity index is 0.70-0.91 (Squires et al., 2013)。

CONTACTS AND LOCATIONS:
Overall Officials: Hao-Yuan Chang, Asst. Prof., Study Chair — School of Nursing, College of Medicine, National Taiwan University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yeh, W. Y., Cheng, Y. W., Chen, M. J., Chiu, H. W. (2008). Development and validation of an occupational burnout inventory. Taiwan Journal of Public Health, 27(5)，349-464.
- [Background] Yang, W. C., Hu, C. H., Wu, I, T. (2014). This study the relationship of working hours, stress studies and workplace fatigue in nursing staff. Journal of Sport and Recreation Management, 11 (1), 114-131.
- [Background] Bagley CL, Rendas-Baum R, Maglinte GA, Yang M, Varon SF, Lee J, Kosinski M. Validating Migraine-Specific Quality of Life Questionnaire v2.1 in episodic and chronic migraine. Headache. 2012 Mar;52(3):409-21. doi: 10.1111/j.1526-4610.2011.01997.x. Epub 2011 Sep 19. PMID 21929662
- [Background] French DJ, Holroyd KA, Pinell C, Malinoski PT, O'Donnell F, Hill KR. Perceived self-efficacy and headache-related disability. Headache. 2000 Sep;40(8):647-56. doi: 10.1046/j.1526-4610.2000.040008647.x. PMID 10971661
- [Background] Lovibond, S. H., & Lovibond, P. F.(2004). Manual for the depression anxiety stress scale. (2nd Ed.). Sydney, Australia: Psychology Foundation Monograph.
- [Background] Mason, M. (1996). Aromatherapy and midwifery. Aromatherapy. Quarterly spring issue, 32-34.
- [Background] Melzack R. The McGill Pain Questionnaire: major properties and scoring methods. Pain. 1975 Sep;1(3):277-299. doi: 10.1016/0304-3959(75)90044-5. PMID 1235985
- [Background] Moussa, M.T., Lovibond, P.F. & Laube, R. (2001). Psychometric properties of a Chinese version of the short Depression Anxiety Stress Scales (DASS21). Report for New South Wales Transcultural Mental Health Centre, Cumberland Hospital, Sydney.
- [Background] Teng CI, Lotus Shyu YI, Chang HY. Moderating effects of professional commitment on hospital nurses in Taiwan. J Prof Nurs. 2007 Jan-Feb;23(1):47-54. doi: 10.1016/j.profnurs.2006.10.002. PMID 17292133
- [Background] Aiken LH, Clarke SP, Sloane DM, Sochalski JA, Busse R, Clarke H, Giovannetti P, Hunt J, Rafferty AM, Shamian J. Nurses' reports on hospital care in five countries. Health Aff (Millwood). 2001 May-Jun;20(3):43-53. doi: 10.1377/hlthaff.20.3.43. PMID 11585181
- [Background] Ball JE, Murrells T, Rafferty AM, Morrow E, Griffiths P. 'Care left undone' during nursing shifts: associations with workload and perceived quality of care. BMJ Qual Saf. 2014 Feb;23(2):116-25. doi: 10.1136/bmjqs-2012-001767. Epub 2013 Jul 29. PMID 23898215
- [Background] Lucero RJ, Lake ET, Aiken LH. Variations in nursing care quality across hospitals. J Adv Nurs. 2009 Nov;65(11):2299-310. doi: 10.1111/j.1365-2648.2009.05090.x. Epub 2009 Sep 8. PMID 19737326
- [Background] Schubert M, Glass TR, Clarke SP, Schaffert-Witvliet B, De Geest S. Validation of the Basel Extent of Rationing of Nursing Care instrument. Nurs Res. 2007 Nov-Dec;56(6):416-24. doi: 10.1097/01.NNR.0000299853.52429.62. PMID 18004188
- [Background] Squires A, Aiken LH, van den Heede K, Sermeus W, Bruyneel L, Lindqvist R, Schoonhoven L, Stromseng I, Busse R, Brzostek T, Ensio A, Moreno-Casbas M, Rafferty AM, Schubert M, Zikos D, Matthews A. A systematic survey instrument translation process for multi-country, comparative health workforce studies. Int J Nurs Stud. 2013 Feb;50(2):264-73. doi: 10.1016/j.ijnurstu.2012.02.015. Epub 2012 Mar 23. PMID 22445444